CLINICAL TRIAL: NCT02412059
Title: Topical Use of Corticosteroid to Prevent Epiretinal Membrane Formation in Eyes With Retinal Tear Undergoing Laser Retinopexy: a Pilot Prospective Clinical Study
Brief Title: Topical Use of Corticosteroid to Prevent Epiretinal Membrane Following Retinal Tear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: LichterM
Record Dates: First submitted 2015-04-03; First posted 2015-04-08 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Epiretinal Membrane
MeSH Terms: conditions — Epiretinal Membrane | interventions — prednisolone acetate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prednisolone (Experimental): Pred Forte (prednisolone acetate ophthalmic suspension, USP) 1% sterile
  Interventions: Drug: Prednisolone acetate
- Control (No Intervention): Patients in control group will not be given a corticosteroid as per usual standard of care.

INTERVENTIONS:
Drug: Prednisolone acetate
  Other Names: Pred Forte
  Arms: Prednisolone

SUMMARY:
In this prospective randomized controlled double blind pilot clinical study, we aim to assess whether administration of a topical corticosteroid would attenuate epiretinal membrane formation following development of retinal tears treated with laser retionpexy.

DETAILED DESCRIPTION:
Epiretinal membrane (ERM) is a frequent, sight-threatening eye condition occurring in 1.02% - 28.9% of eyes in persons aged 40 years or older. [1] While often idiopathic in nature, ERM formation has been associated with retinal tears, possibly due to a breakdown of the blood-retinal barrier [1-3]. Pathological analysis of ERM content shows inflammatory mediators such as cytokines, growth factors and interleukins, which can promote fibroblast remodelling that leads to a contractile scar formation on the retinal surface. [1, 4-8] For this reason, ERM formation has been suggested to be an aberrant tissue repair or wound-healing process driven by inflammatory reactions. Since corticosteroids inhibit the inflammatory cascade and fibroblast transdifferentiation, administration of a corticosteroid following retinal tears should theoretically reduce the risk of ERM formation. [9-10] In this study, we aim to assess whether administration of a topical corticosteroid would attenuate ERM formation following laser retinopexy of retinal tears.

ELIGIBILITY:
Inclusion Criteria:

* Between ages 18 to 80 (inclusive)
* English-speaking
* Undergoing non-pneumatic laser retinopexy procedure for horseshoe retinal tear (without retinal detachment)

Exclusion Criteria:

* Patient refusal or delay of retinopexy procedure for more than 48 hours after diagnosis
* Patients who are pseudophakic or aphakic
* Medical conditions contraindicated with prednisolone: viral diseases of the cornea and conjunctiva including herpes simplex, vaccinia, varicella; fundal diseases of ocular structures; mycobacterial infections; hypercortisolism.
* Previous history of epiretinal membrane, retinal surgery (cryo or laser)
* Patients with hypersensitivity or contraindication for corticosteroids (viral diseases of the cornea and conjunctiva including herpes simplex, vaccinia, varicella; fungal diseases of ocular structures; mycobacterial infections; hypercortisolism).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-08; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Incidence of epiretinal membrane | 6-months following administration of corticosteroid

CONTACTS AND LOCATIONS:
Overall Officials: Myrna Lichter, MD, FRCSC, Principal Investigator — University of Toronto Department of Ophthalmology

REFERENCES:
- [Background] Bu SC, Kuijer R, Li XR, Hooymans JM, Los LI. Idiopathic epiretinal membrane. Retina. 2014 Dec;34(12):2317-35. doi: 10.1097/IAE.0000000000000349. PMID 25360790
- [Background] Saran BR, Brucker AJ. Macular epiretinal membrane formation and treated retinal breaks. Am J Ophthalmol. 1995 Oct;120(4):480-5. doi: 10.1016/s0002-9394(14)72662-5. PMID 7573306
- [Background] Snead DR, James S, Snead MP. Pathological changes in the vitreoretinal junction 1: epiretinal membrane formation. Eye (Lond). 2008 Oct;22(10):1310-7. doi: 10.1038/eye.2008.36. Epub 2008 Mar 14. PMID 18344963
- [Background] Joshi M, Agrawal S, Christoforidis JB. Inflammatory mechanisms of idiopathic epiretinal membrane formation. Mediators Inflamm. 2013;2013:192582. doi: 10.1155/2013/192582. Epub 2013 Nov 11. PMID 24324293
- [Background] Gilbert C, Hiscott P, Unger W, Grierson I, McLeod D. Inflammation and the formation of epiretinal membranes. Eye (Lond). 1988;2 Suppl:S140-56. doi: 10.1038/eye.1988.140. PMID 3076143
- [Background] Hiscott PS, Unger WG, Grierson I, McLeod D. The role of inflammation in the development of epiretinal membranes. Curr Eye Res. 1988 Sep;7(9):877-92. doi: 10.3109/02713688808997245. PMID 3180837
- [Background] Grinnell F. Fibroblasts, myofibroblasts, and wound contraction. J Cell Biol. 1994 Feb;124(4):401-4. doi: 10.1083/jcb.124.4.401. No abstract available. PMID 8106541
- [Background] Banerjee PJ, Woodcock MG, Bunce C, Scott R, Charteris DG. A pilot study of intraocular use of intensive anti-inflammatory; triamcinolone acetonide to prevent proliferative vitreoretinopathy in eyes undergoing vitreoretinal surgery for open globe trauma; the Adjuncts in Ocular Trauma (AOT) Trial: study protocol for a randomised controlled trial. Trials. 2013 Feb 13;14:42. doi: 10.1186/1745-6215-14-42. PMID 23406256
- [Background] Tano Y, Sugita G, Abrams G, Machemer R. Inhibition of intraocular proliferations with intravitreal corticosteroids. Am J Ophthalmol. 1980 Jan;89(1):131-6. doi: 10.1016/0002-9394(80)90239-1. PMID 6153251